CLINICAL TRIAL: NCT05598710
Title: Ureteral Stent Related Lower Urinary Tract Symptoms- A Comparative Study
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Bellos Themistoklis, Urology Intern, National and Kapodistrian University of Athens
Other Study IDs: 14778
Record Dates: First submitted 2022-10-25; First posted 2022-10-28 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Ureteral Stent-Related Symptom
Keywords: pigtail; ureteral stent; USSQ; pigtail size; pigtail length; LUTS; hematuria; pain; sexual performance; daily activity; professional performance
MeSH Terms: conditions — Hematuria; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Group who have pigtail 5-26
  Interventions: Procedure: Pigtail Insertion
- Group 2: Group who have pigtail 6-26
  Interventions: Procedure: Pigtail Insertion
- Group 3: Group who have pigtail 5-28
  Interventions: Procedure: Pigtail Insertion
- Group 4: Group who have pigtail 6-28
  Interventions: Procedure: Pigtail Insertion

INTERVENTIONS:
Procedure: Pigtail Insertion — Pigtail is inserted for any reason of ureteral obstruction except for malignant

SUMMARY:
Pigtails are inserted to relieve of pelviureteral system independent of the underlying cause. Pain, Lower Urinary Tract Symptoms (LUTS), hematuria and fever can be some of the early complications after their insertion..More than 80% of the patients mention significant amount of pain limiting their daily activities while 78% mentions LUTS.

The local irritation from the pigtail in the kidney and the ureterovesical junction, the urine reflux through the pigtail, length and size of the pigtail are some of the factors that account for the Ureteral Stent Related Symptoms (USRS) .Important role also has the length of remaining pigtail within the bladder as well as the drainage capacity,the lack of elasticity and the migration within the bladder of the pigtail .Aim of this study is to correlate the physical properties of the pigtail (length,size) with the complications after the insertion.

DETAILED DESCRIPTION:
Ureteral stents were first described by Finney and Hepperlen. Stenting of the upper urinary tract was initially used for relieving upper urinary tract obstruction and for ureteral alignment. The first self retaining ureteral catheters were described by Gibbons , Mardis , Finney and Hepperlen. Ureteral stents can be either open -end or close- end. The main materials used for manufacturing them are silicone, polyurethane and Percuflex.

Pigtail are placed to prevent ureteral obstruction from stone fragments, ureteral oedema, hepatoma, as well as to prevent urinomas.Some of the factors that influence Ureteral Stent Related Symptoms ( USSQ) are the irritation to the kidney and bladder trigone, the vesicoureteral reflux through the pigtail ,pigtail length and the remaining tail length within the bladder.Early complications after pigtail insertion include pain, LUTS (lower urinary tract symptoms )[ increased frequency (60%), hesitancy (60%) ,dysuria (40%)] , renal pain ,body pain, hematuria (54%) and fever. More than 80% of the patients mention pain limiting their daily activities while 78% mentions LUTS. Late complications following pigtail insertion include pigtail migration , renal obstruction , stone formation around the pigtail and automatic pigtail degradation.Pigtail can also affect sexual and professional life.

The purpose of this survey is to clarify the connection between the pigtail physical properties (length, size) with the complications arising from their use.The goal is to investigate if the use of one type of ureteral stent with particular characteristics is better than the others and the use of this knowledge in everyday clinical praxis.

In this survey will be included patients with inserted pigtails. In our clinic we have access to pigtail sizes 6 Fr 26 cm, 5 Fr 26 cm,6 Fr 28 cm και 5 Fr 28 cm.The patients will be divided into 4 groups depending on the pigtail size. All the patients will have signed a consent form prior to their inclusion in the study. Patients having pigtail due to malignant disease and patients not being in the mental state to cooperate will be excluded from this survey. The pigtail insertion will be correlated with the potential complications using the Ureteral Stent Related Symptoms Questionnaire ( USSQ) which was first described by Joshi in 2003. This questionnaire is answered by each patient the first and fourth week of pigtail insertion and the fourth week after pigtail removal. It includes questions covering six fields: urinary tract symptoms, body pain, overall health, professional performance , sexual performance and additional problems.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inserted pigtails

Exclusion Criteria:

* Mental disorder
* Ureteral obstruction due to malignant disease
* Patients with LUTS due to benign prostatic hyperplasia(BPH)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inserted pigtails due to ureteral obstruction or due to procedures such as URS, RIRS and PCNL
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Correlation of Ureteral Stent related symptoms with pigtail physical characteristics | 2 years
  Correlation of Ureteral Stent related symptoms with pigtail physical characteristics

SECONDARY OUTCOMES:
Correlation of Ureteral Stent related symptoms with patients characteristics (height) | 2 years
  Correlation of Ureteral Stent related symptoms with patients characteristics (height)

CONTACTS AND LOCATIONS:
Locations (1):
- Themistoklis Bellos, Marathon, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finney RP. Experience with new double J ureteral catheter stent. J Urol. 1978 Dec;120(6):678-81. doi: 10.1016/s0022-5347(17)57326-7. PMID 731804
- [Result] Beiko DT, Knudsen BE, Denstedt JD. Advances in ureteral stent design. J Endourol. 2003 May;17(4):195-9. doi: 10.1089/089277903765444294. PMID 12816579
- [Result] Hepperlen TW, Mardis HK, Kammandel H. Self-retained internal ureteral stents: a new approach. J Urol. 1978 Jun;119(6):731-4. doi: 10.1016/s0022-5347(17)57613-2. PMID 77917
- [Result] Gibbons RP, Mason JT, Correa RJ Jr. Experience with indwelling silicone rubber ureteral catheters. J Urol. 1974 May;111(5):594-9. doi: 10.1016/s0022-5347(17)60023-5. No abstract available. PMID 4823967
- [Result] Mardis HK, Hepperlen TW, Kammandel H. Double pigtail ureteral stent. Urology. 1979 Jul;14(1):23-6. doi: 10.1016/0090-4295(79)90205-x. PMID 452213
- [Result] Lam JS, Gupta M. Tips and tricks for the management of retained ureteral stents. J Endourol. 2002 Dec;16(10):733-41. doi: 10.1089/08927790260472881. PMID 12542876
- [Result] Dellis A, Joshi HB, Timoney AG, Keeley FX Jr. Relief of stent related symptoms: review of engineering and pharmacological solutions. J Urol. 2010 Oct;184(4):1267-72. doi: 10.1016/j.juro.2010.06.043. Epub 2010 Aug 17. PMID 20723923
- [Result] Liu Q, Liao B, Zhang R, Jin T, Zhou L, Luo D, Liu J, Li H, Wang K. Combination therapy only shows short-term superiority over monotherapy on ureteral stent-related symptoms - outcome from a randomized controlled trial. BMC Urol. 2016 Nov 15;16(1):66. doi: 10.1186/s12894-016-0186-y. PMID 27846839
- [Result] Giannarini G, Keeley FX Jr, Valent F, Manassero F, Mogorovich A, Autorino R, Selli C. Predictors of morbidity in patients with indwelling ureteric stents: results of a prospective study using the validated Ureteric Stent Symptoms Questionnaire. BJU Int. 2011 Feb;107(4):648-54. doi: 10.1111/j.1464-410X.2010.09482.x. PMID 20590539
- [Result] Cubuk A, Yanaral F, Ozgor F, Savun M, Ozdemir H, Erbin A, Yuksel B, Sarilar O. Comparison of 4.8 Fr and 6 Fr ureteral stents on stent related symptoms following ureterorenoscopy: A prospective randomized controlled trial. Kaohsiung J Med Sci. 2018 Dec;34(12):695-699. doi: 10.1016/j.kjms.2018.07.001. Epub 2018 Jul 21. PMID 30527204
- [Result] Thomas R. Indwelling ureteral stents: impact of material and shape on patient comfort. J Endourol. 1993 Apr;7(2):137-40. doi: 10.1089/end.1993.7.137. PMID 8518826
- [Result] Ahallal Y, Khallouk A, El Fassi MJ, Farih MH. Risk factor analysis and management of ureteral double-j stent complications. Rev Urol. 2010 Spring;12(2-3):e147-51. PMID 20811552
- [Result] Betschart P, Zumstein V, Piller A, Schmid HP, Abt D. Prevention and treatment of symptoms associated with indwelling ureteral stents: A systematic review. Int J Urol. 2017 Apr;24(4):250-259. doi: 10.1111/iju.13311. Epub 2017 Feb 25. PMID 28236323